CLINICAL TRIAL: NCT05197673
Title: Identifying Risks of Outbreaks in Work Settings and the Implications for Control Measures
Brief Title: Identifying Risks of COVID-19 Outbreaks in Work Settings and the Implications for Control Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tse Lap Ah, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021.531-T
Record Dates: First submitted 2021-11-30; First posted 2022-01-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Intention to Get SARS-CoV-2 Vaccination; Intention to Get SARS-CoV-2 Antibody Test
Keywords: workplace hazards; exposure prevention; vaccination; SARS-CoV-2; control measures; willingness; attitude; antibody testing
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Intervention group will receive theory-based educational intervention using the Theory of Planned Behaviours (TPB) PLUS general health information; Control group will receive only general health information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This arm will receive TPB intervention to build positive attitudes towards COVID-19 related preventive behaviour (e.g., good compliance with infection control measures, encouraging uptake of testing and vaccination), subjective norms (tackling strategies for perceived social pressure from others or normative beliefs), and improve perceived behavioural control towards risks of outbreaks in workplace.
  Interventions: Behavioral: Theory of planned behaviours (TPB) based intervention
- Control group (No Intervention): Control group will receive only general health information.

INTERVENTIONS:
Behavioral: Theory of planned behaviours (TPB) based intervention — Intervention group will receive TPB-based education program to improve workers' attitude toward SARS-CoV-2 and raise their intention to vaccination and virus testing. The intervention will be implemented at the baseline with measurements repeated at the 3rd month, 6th month and 9th month. The standardized mode of intervention includes face-to-face/online seminar (depends on the COVID-19 situation), message via mobile phone, promotion pamphlet, etc.
  Arms: Intervention group

SUMMARY:
Objectives: To identify core and cross-time workplace hazards and worker's exposure prevention profile towards outbreaks in three non-healthcare work settings; to evaluate effectiveness of a theory-based educational programme on improving attitude to vaccination and virus testing in workplace; to longitudinally compare attitude of willingness to vaccination, testing of SARS-CoV-2 and changes of risk profile toward outbreaks among workers.

Design: A 5-year study comprising a randomized controlled trial (RCT) and 3 parallel longitudinal studies with baseline and follow-up repeated measurements.

Setting: Non-office, mobile and office work settings. Participants: Part I is a RCT, 294 workers will be randomised to an intervention group (a theory-based education programme) and a control group with measurements repeated at 3rd, 6th and 9th month. Part II is a longitudinal quantitative study (i.e., prospective cohort study) involving 1,495 workers recruited at the baseline and followed up for 2 years. Part III is a longitudinal qualitative study involving 26 management and frontline workers. Part IV is a longitudinal workplace hygiene study involving 6 workplaces enrolled at the baseline and followed up to conduct ventilation investigation.

Intervention: Theory-based education intervention to build positive attitude of control measures towards SARS-CoV-2 outbreak.

Main outcome measure: Workplace hygiene data (airflow, air volume, etc.); willingness to vaccination and virus tests; actual uptake of SARS-CoV-2 antibody testing.

Data analyses: Multivariate regression logistic model and thematically analysed will be performed for quantitative and qualitative analysis. Intention-to-treat analysis will be employed for RCT.

Expected results: Large dataset of longitudinal measurement of willingness to vaccination/testing and actual uptake will be documented to inform policy. Educational intervention will be developed to mitigate risks of outbreaks in workplace.

ELIGIBILITY:
Inclusion Criteria:

* currently being employed in Hong Kong

Exclusion Criteria:

* who have history of physician-diagnosed cancer and sever chronic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change of intention to get vaccination of SARS-CoV-2 | 3rd, 6th and 9th month
  A questionnaire will be used to evaluate the intention to get vaccination quantitively. This assessment will be repeated in the 3rd, 6th and 9th month. Change will be assessed among these time points.

SECONDARY OUTCOMES:
Change of intention to uptake SARS-CoV-2 antibody test | 3rd, 6th and 9th month
  A questionnaire will be used to evaluate the intention to get rapid antibody test quantitively. This assessment will be repeated in the 3rd, 6th and 9th month. Change will be assessed among these time points.

CONTACTS AND LOCATIONS:
Overall Officials: Lap Ah Tse, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

REFERENCES:
- [Derived] Tse LA, Wang F, Mo PKH, Wan CCM, Tang NHY, Yang S, Dong D, Ho KF, Wong SY. Does enhanced educational intervention reduce breakthrough infection and mental health problems via improving acceptance of COVID-19 booster shots in Chinese non-healthcare workers: A randomized controlled trial? J Infect Public Health. 2025 May;18(5):102719. doi: 10.1016/j.jiph.2025.102719. Epub 2025 Feb 21. PMID 40056893
- [Derived] Constantin AM, Noertjojo K, Sommer I, Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, McElvenny DM, Rhodes S, Martin C, Sampson O, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD015112. doi: 10.1002/14651858.CD015112.pub3. PMID 38597249

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT05197673/Prot_SAP_000.pdf